CLINICAL TRIAL: NCT00400764
Title: A Phase Ib/II, Open-Label, Multicenter Study of the Safety, Pharmacokinetics, and Efficacy of Dulanermin Administered Intravenously in Combination With Rituximab to Subjects With Follicular and Other Low-Grade, CD20+, B-Cell Non-Hodgkin's Lymphomas That Have Progressed Following Previous Rituximab Therapy
Brief Title: A Study of Dulanermin in Combination With Rituximab in Subjects With Follicular and Other Low Grade, CD20+, Non-Hodgkin's Lymphomas
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APO3585g
Record Dates: First submitted 2006-11-15; First posted 2006-11-17 (Estimated); Results first posted 2011-10-07 (Estimated); Last update posted 2011-11-23 (Estimated); Status verified 2011-11

CONDITIONS: Non-Hodgkin's Lymphoma
Keywords: NHL; Follicular NHL; Rituxan; Apo2L/TRAIL
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — TNFSF10 protein, human; Rituximab

ARMS (5):
- Phase Ib: Dulanermin 4 mg/kg (Experimental): Participants received 4.0 mg/kg/day dose of dulanermin, administered by intravenous (IV) infusion for 5 consecutive days at the start of each 21-day treatment cycle for up to four cycles. Participants also received rituximab administered by IV infusion at 375 mg/m^2 weekly for up to eight doses.
  Interventions: Drug: Dulanermin; Drug: Rituximab
- Phase Ib: Dulanermin 8 mg/kg (Experimental): Participants received 8.0 mg/kg/day dose of dulanermin, administered by intravenous (IV) infusion for 5 consecutive days at the start of each 21-day treatment cycle for up to four cycles. Participants also received rituximab administered by IV infusion at 375 mg/m^2 weekly for up to eight doses.
  Interventions: Drug: Dulanermin; Drug: Rituximab
- Phase II: Rituximab (Active Comparator): Participants received rituximab administered by intravenous (IV) infusion at 375 mg/m^2 weekly for up to eight doses.
  Interventions: Drug: Rituximab
- Phase II: Combination Therapy (Experimental): Participants received 8.0 mg/kg/day dose of dulanermin, administered by intravenous (IV) infusion for 5 consecutive days at the start of each 21-day treatment cycle for up to four cycles. Participants also received rituximab administered by IV infusion at 375 mg/m^2 weekly for up to eight doses.
  Interventions: Drug: Dulanermin; Drug: Rituximab
- Phase II: Dulanermin (Experimental): Participants received 8.0 mg/kg/day dose of dulanermin, administered by intravenous (IV) infusion for 5 consecutive days at the start of each 21-day treatment cycle for up to four cycles.
  Interventions: Drug: Dulanermin

INTERVENTIONS:
Drug: Dulanermin — Dulanermin was administered by intravenous (IV) infusion over 1 hour on days 1-5 of each 21-day cycle.
  Arms: Phase II: Combination Therapy; Phase II: Dulanermin; Phase Ib: Dulanermin 4 mg/kg; Phase Ib: Dulanermin 8 mg/kg
Drug: Rituximab — Rituximab was administered by intravenous (IV) infusion at 375 mg/m^2 weekly for up to eight doses.
  Arms: Phase II: Combination Therapy; Phase II: Rituximab; Phase Ib: Dulanermin 4 mg/kg; Phase Ib: Dulanermin 8 mg/kg

SUMMARY:
This Phase Ib/II, open-label, multicenter trial is designed to evaluate the safety, pharmacokinetics, and efficacy of dulanermin when combined with rituximab in subjects with follicular, CD20+, B-cell Non-Hodgkin's Lymphoma (NHL) that has progressed following a response of ≥ 6 months duration to a prior rituximab-containing therapy. The multicenter, international, randomized Phase II part of this study will commence only after the safety and available pharmacokinetic data from the Phase Ib part of the study have been evaluated by the Sponsor and have been provided to participating investigators and the FDA.

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent Form
* Age ≥ 18 years
* History of histologically confirmed CD20+ follicular NHL Grade 1, 2, or 3a
* Progression of disease following the most recent treatment with rituximab-containing therapy that resulted in stable disease or a partial or complete response lasting ≥ 6 months
* Measurable disease
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* For subjects of reproductive potential (males and females), use of a reliable means of contraception (e.g., contraceptive pill, intrauterine device [IUD], physical barrier throughout the trial and for 1 year following their final exposure to study treatment).
* Life expectancy of > 3 months

Exclusion Criteria:

* Prior radiotherapy to a measurable, metastatic lesion(s) to be used to measure response unless that lesion shows unequivocal progression at baseline
* Radiation therapy to a peripheral lesion within 14 days prior to Day 1; Radiation therapy to a thoracic, abdominal, or pelvic field within 28 days prior to Day 1
* Chemotherapy, hormonal therapy, radiotherapy, or immunotherapy within 4 weeks prior to Day 1
* Patients who have received radioimmunotherapy for relapsed or refractory, follicular NHL are eligible for the study if they received this therapy at least 1 year prior to Day 1, they have adequate bone marrow function, and they have no evidence of myelodysplastic syndrome on bone marrow aspirate/biopsy
* Prior treatment with dulanermin or an agonist antibody to DR4 or DR5
* Concurrent systemic corticosteroid therapy
* Evidence of clinically detectable ascites on Day 1
* Other invasive malignancies within 5 years prior to Day 1
* History or evidence upon physical examination of central nervous system (CNS) disease within 1 year prior to study entry
* Active infection requiring parenteral antibiotics on Day 1
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to Day 1 or anticipation of need for major surgical procedure during the course of the study and fine needle aspirations within 7 days prior to Day 1
* Pregnancy or lactation
* Serious nonhealing wound, ulcer, or bone fracture
* Current or recent participation in another experimental drug study
* Clinically significant cardiovascular disease
* Known positive test result for HIV, hepatitis B surface antigen (sAg), hepatitis B IgG or IgM core antibody, or hepatitis C antibody
* Known sensitivity to murine or human antibodies
* History of other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates use of an investigational drug or that might affect interpretation of the results of the study or render the subject at high risk from treatment complications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2006-06; Primary Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chia Portera, PhD., M.D, Study Director — Genentech, Inc.

REFERENCES:
- [Derived] Cheah CY, Belada D, Fanale MA, Janikova A, Czucman MS, Flinn IW, Kapp AV, Ashkenazi A, Kelley S, Bray GL, Holden S, Seymour JF. Dulanermin with rituximab in patients with relapsed indolent B-cell lymphoma: an open-label phase 1b/2 randomised study. Lancet Haematol. 2015 Apr;2(4):e166-74. doi: 10.1016/S2352-3026(15)00026-5. Epub 2015 Mar 25. PMID 26687959

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The Phase Ib part of this study was completed prior to the start of Phase II. Phase Ib participants were not eligible for participation in Phase II.
Groups:
- Phase Ib - Dulanermin 4 mg/kg: Participants received 4.0 mg/kg/day dose of dulanermin, administered by intravenous (IV) infusion for 5 consecutive days at the start of each 21-day treatment cycle for up to four cycles. Participants also received rituximab administered by IV infusion at 375 mg/m^2 weekly for up to eight doses.
- Phase Ib - Dulanermin 8 mg/kg; Phase II - Combination Therapy: Participants received 8.0 mg/kg/day dose of dulanermin, administered by intravenous (IV) infusion for 5 consecutive days at the start of each 21-day treatment cycle for up to four cycles. Participants also received rituximab administered by IV infusion at 375 mg/m^2 weekly for up to eight doses.
- Phase II - Rituximab: Participants received rituximab administered by intravenous (IV) infusion at 375 mg/m^2 weekly for up to eight doses.
- Phase II - Dulanermin: Participants received 8.0 mg/kg/day dose of dulanermin, administered by intravenous (IV) infusion for 5 consecutive days at the start of each 21-day treatment cycle for up to four cycles.
Period: Phase Ib
Arm/Group | Phase Ib - Dulanermin 4 mg/kg | Phase Ib - Dulanermin 8 mg/kg | Phase II - Rituximab | Phase II - Combination Therapy | Phase II - Dulanermin
Started | 6 | 6 | 0 | 0 | 0
Treated | 6 | 6 | 0 | 0 | 0
Completed | 0 (One patient reported as discontinued due to an AE should have been reported as death.) | 2 | 0 | 0 | 0
Not Completed | 6 | 4 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0 | 0
Not completed — Death | 1 | 0 | 0 | 0 | 0
Not completed — Disease Progression | 4 | 4 | 0 | 0 | 0
Period: Phase II
Arm/Group | Phase Ib - Dulanermin 4 mg/kg | Phase Ib - Dulanermin 8 mg/kg | Phase II - Rituximab | Phase II - Combination Therapy | Phase II - Dulanermin
Started | 0 | 0 | 23 | 26 | 11
Treated | 0 | 0 | 22 (One patient in the Rituximab arm withdrew prior to treatment) | 26 | 11
Completed | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 23 | 26 | 11
Not completed — Death | 0 | 0 | 1 | 2 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 1 | 1 | 0
Not completed — Sponsor's decision to terminate | 0 | 0 | 18 | 22 | 11
Not completed — Patient began new, non-protocol, therapy | 0 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase Ib - Dulanermin 4 mg/kg | Phase Ib - Dulanermin 8 mg/kg | Phase II - Rituximab | Phase II - Combination Therapy | Phase II - Dulanermin | Total
Number analyzed (Participants) | 6 | 6 | 22 | 26 | 11 | 71
Age Continuous [Mean (Standard Deviation); unit: years] — Age demographic data for the Phase Ib population.
  years | 56.3 (15.9) | 63.7 (9.0) | NA (NA) — Age demographic data for the Phase Ib population. | NA (NA) — Age demographic data for the Phase Ib population. | NA (NA) — Age demographic data for the Phase Ib population. | 60.0 (12.9)
Age, Customized [Mean (Standard Deviation); unit: years] — Age demographic data for the Phase II population.
  years | NA (NA) — Age demographic data for the Phase II population. | NA (NA) — Age demographic data for the Phase II population. | 58.0 (8.5) | 58.4 (9.8) | 61.4 (13.3) | 58.8 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 9 | 7 | 2 | 20
  Male | 5 | 5 | 13 | 19 | 9 | 51

OUTCOME MEASURES:

1. Primary Outcome: Phase Ib: Number of Participants With a Dose-limiting Toxicity
Description: A dose-limiting toxicity (DLT) was defined as a National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v3.0 Grade ≥ 3 hematologic or major organ toxicity that was related to study drug (i.e., dulanermin). Although a patient may have experienced a DLT at any time during the study, only events that occurred within the DLT assessment window were considered for dose-escalation decisions and determination of the maximum tolerated dose (MTD).
Time Frame: The DLT assessment window was defined as the duration required to complete two full cycles of treatment with dulanermin (2 * 21 days) and four doses of rituximab (usually through Day 28).
Population: The DLT-evaluable population consisted of all patients enrolled in the Phase Ib who received at least two complete cycles of dulanermin and four doses of rituximab and complete study assessments through the DLT Assessment Window without a DLT (usually through Day 28) or experienced a DLT and withdrew from the study within the DLT Assessment Window.
Measure: Number; unit: participants
Arm/Group | Phase Ib - Dulanermin 4 mg/kg | Phase Ib - Dulanermin 8 mg/kg
Number analyzed (Participants) | 6 | 6
participants | 0 | 0

2. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events by Severity Grade
Description: Safety was assessed through summaries of treatment-emergent adverse events (AEs); AEs were graded using the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 3.0, according to the following guidelines: Grade 1 (Mild); Grade 2 (Moderate); Grade 3 (Severe); Grade 4 (Life-threatening or disabling) and Grade 5 (Death related to AE).
Time Frame: From Baseline through Study Termination (up to a maximum of approximately 13 months for phase Ib and up to approximately 33 months for phase II)
Population: Safety Evaluable population, consisting of all randomized patients who received at least one dose of treatment.
Measure: Number; unit: participants
Arm/Group | Phase Ib - Dulanermin 4 mg/kg | Phase Ib - Dulanermin 8 mg/kg | Phase II - Rituximab | Phase II - Combination Therapy | Phase II - Dulanermin
Number analyzed (Participants) | 6 | 6 | 22 | 26 | 11
participants
  Grade 5 AE | 0 | 0 | 1 | 0 | 0
  Grade 4 AE | 1 | 0 | 0 | 0 | 0
  Grade 3 AE | 1 | 3 | 1 | 6 | 0
  Grade 2 AE | 4 | 1 | 8 | 10 | 4
  Grade 1 AE | 0 | 2 | 6 | 7 | 4
  Any Grade AEs | 6 | 6 | 16 | 23 | 8

3. Primary Outcome: Phase II: Objective Response as Assessed by the Independent Review Facility (IRF)
Description: Objective response was defined as a confirmed or unconfirmed complete response (CR, CRu) or partial response (PR) assessed on the basis of clinical, radiographic (computed tomography (CT) scans of the neck, chest, abdomen, pelvis and inguinal region), and pathologic (i.e., bone marrow) criteria and according to the modified International Working Group (IWG) criteria. All radiographic and clinical data for the evaluation of objective response were submitted to an IRF for blinded and impartial assessment.
  Patients without a post-baseline tumor assessment were considered non-responders.
Time Frame: From Baseline through Study Termination (up to approximately 33 months)
Population: The phase II Efficacy-Evaluable population consisted of all randomized patients who received at least one dose of study treatment and had measurable disease at baseline, as assessed by the IRF.
Measure: Number; unit: participants
Groups:
- Rituximab: Participants received rituximab administered by intravenous (IV) infusion at 375 mg/m^2 weekly for up to eight doses.
- Combination Therapy: Participants received 8.0 mg/kg/day dose of dulanermin, administered by intravenous (IV) infusion for 5 consecutive days at the start of each 21-day treatment cycle for up to four cycles. Participants also received rituximab administered by IV infusion at 375 mg/m^2 weekly for up to eight doses.
- Dulanermin: Participants received 8.0 mg/kg/day dose of dulanermin, administered by intravenous (IV) infusion for 5 consecutive days at the start of each 21-day treatment cycle for up to four cycles.
Arm/Group | Rituximab | Combination Therapy | Dulanermin
Number analyzed (Participants) | 22 | 25 | 11
participants
  Total Objective Response | 14 | 16 | 1
  Complete Response | 5 | 3 | 0
  Complete Response unconfirmed | 0 | 2 | 0
  Partial Response | 9 | 11 | 1

4. Primary Outcome: Vital Signs: Change From Baseline in Diastolic and Systolic Blood Pressure at Treatment Termination Visit
Description: Blood pressure was measured at baseline and throughout the study. Change from baseline was calculated using the patient's last recorded measurement at the completion of treatment visit - baseline measurement.
Time Frame: Baseline and Treatment Termination visit (8 weeks for Rituximab arm and 12 weeks for combination and Dulanermin arms)
Population: Safety Evaluable population, consisting of all randomized patients who received at least one dose of treatment.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Phase Ib - Dulanermin 4 mg/kg | Phase Ib - Dulanermin 8 mg/kg | Phase II - Rituximab | Phase II - Combination Therapy | Phase II - Dulanermin
Number analyzed (Participants) | 6 | 6 | 22 | 26 | 11
mmHg
  Diastolic Blood Pressure | -8.7 (10.9) | -5.2 (7.9) | 2.3 (9.9) | 1.6 (9.2) | -0.8 (5.6)
  Systolic Blood Pressure | -3.2 (16.8) | -4.7 (10.9) | -3.4 (14.8) | -2.2 (19.6) | -4.2 (9.5)

5. Primary Outcome: Vital Signs: Change From Baseline in Heart Rate at Treatment Termination Visit
Description: Heart rate was measured at baseline and throughout the study. Change from baseline was calculated using the patient's last recorded measurement at the completion of treatment visit - baseline measurement.
Time Frame: Baseline and Treatment Termination visit (8 weeks for Rituximab arm and 12 weeks for combination and Dulanermin arms)
Population: Safety Evaluable population, consisting of all randomized patients who received at least one dose of treatment.
Measure: Mean (Standard Deviation); unit: beats/minute
Arm/Group | Phase Ib - Dulanermin 4 mg/kg | Phase Ib - Dulanermin 8 mg/kg | Phase II - Rituximab | Phase II - Combination Therapy | Phase II - Dulanermin
Number analyzed (Participants) | 6 | 6 | 22 | 26 | 11
beats/minute | 7.0 (21.4) | -1.5 (6.7) | 0.5 (9.6) | 3.3 (10.6) | 5.0 (13.2)

6. Secondary Outcome: Phase II: Progression Free Survival
Description: Progression free survival (PFS) was defined as the time from randomization to documented disease progression or death, whichever occurred first and was based on the investigator's assessment using the modified IWG criteria. Kaplan-Meier methods were used to estimate median time to PFS. Data for patients without disease progression or death on study were censored at the time of the last tumor assessment.
Time Frame: From Baseline through Study Termination (up to approximately 33 months)
Population: Safety-Evaluable population consisting of all randomized patients who received at least one dose of study treatment
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Rituximab | Combination Therapy | Dulanermin
Number analyzed (Participants) | 22 | 26 | 11
months | 29.9 [9.2 to 29.9] | 17.9 [9.9 to 18.4] | 6.9 [2.9 to NA] — The upper limit of the confidence interval was not estimable due to low numbers of events.

7. Secondary Outcome: Phase II: Overall Survival
Description: Median overall survival could not be estimated because of the low number of deaths at the time of study termination.
Time Frame: From Baseline through Study Termination (up to approximately 33 months)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Rituximab | Combination Therapy | Dulanermin
Number analyzed (Participants) | 0 | 0 | 0

8. Secondary Outcome: Phase II: Objective Response as Assessed by the Investigator
Description: Objective response was defined as a confirmed or unconfirmed complete response(CR, CRu) or partial response (PR) assessed on the basis of clinical, radiographic (computed tomography (CT) scans of the neck, chest, abdomen, pelvis and inguinal region), and pathologic (i.e., bone marrow) criteria and according to the modified International Working Group (IWG) criteria. Patients without a post-baseline tumor assessment were considered non-responders.
Time Frame: From Baseline through Study Termination (up to approximately 33 months)
Population: Safety Evaluable population, consisting of all randomized patients who received at least one dose of treatment.
Measure: Number; unit: participants
Arm/Group | Rituximab | Combination Therapy | Dulanermin
Number analyzed (Participants) | 22 | 26 | 11
participants
  Total Objective Response | 15 | 17 | 1
  Complete Response | 7 | 7 | 1
  Complete Response unconfirmed | 0 | 1 | 0
  Partial Response | 8 | 9 | 0

9. Secondary Outcome: Phase II: Duration of Response as Assessed by the Investigator
Description: An event was defined as documented disease progression or death on study, whichever occurred first. Duration of objective response was defined only for patients with an objective response as determined by the investigator and was the time from the initial response to disease progression or death on study.
  Kaplan-Meier methods were used to estimate median, percentiles, and range of duration of response.
Time Frame: From Baseline through Study Termination (up to approximately 33 months)
Population: Safety-evaluable patients with an objective response determined by the Investigator.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Rituximab | Combination Therapy | Dulanermin
Number analyzed (Participants) | 15 | 17 | 1
months | 21.4 [7.7 to 21.4] | 11.3 [8.0 to NA] — Could not be calculated due to low number of patients with events. | NA [NA to NA] — Median duration of objective response could not be estimated for the dulanermin only arm because only 1 patient had an objective response based on investigator assessment

10. Primary Outcome: Vital Signs: Change From Baseline in Body Temperature at Treatment Termination Visit
Description: Body temperature was measured at baseline and throughout the study. Change from baseline was calculated using the patients last recorded measurement at the completion of treatment visit - baseline measurement.
Time Frame: Baseline and Treatment Termination visit (8 weeks for Rituximab arm and 12 weeks for combination and Dulanermin arms)
Population: Safety Evaluable population, consisting of all randomized patients who received at least one dose of treatment.
Measure: Mean (Standard Deviation); unit: degrees Celsius
Arm/Group | Phase Ib - Dulanermin 4 mg/kg | Phase Ib - Dulanermin 8 mg/kg | Phase II - Rituximab | Phase II - Combination Therapy | Phase II - Dulanermin
Number analyzed (Participants) | 6 | 6 | 22 | 26 | 11
degrees Celsius | -0.0 (0.6) | -0.3 (0.7) | 2.8 (13.1) | -0.1 (0.4) | 0.0 (0.4)

11. Primary Outcome: Number of Participants With a Clinically Significant Laboratory Abnormality
Description: Laboratory Parameters were graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE). A clinically significant abnormality was defined as a Grade 3 (severe) or Grade 4 (very severe, life threatening, or disabling) laboratory toxicity according to the NCI CTCAE v3.0.
Time Frame: Baseline and Treatment Termination visit (8 weeks for Rituximab arm and 12 weeks for combination and Dulanermin arms).
Population: Safety Evaluable population consisting of all randomized patients who received at least one dose of study drug.
Measure: Number; unit: participants
Arm/Group | Phase Ib - Dulanermin 4 mg/kg | Phase Ib - Dulanermin 8 mg/kg | Phase II - Rituximab | Phase II - Combination Therapy | Phase II - Dulanermin
Number analyzed (Participants) | 6 | 6 | 22 | 26 | 11
participants | 3 | 4 | 5 | 11 | 5

12. Primary Outcome: Mean Serum Concentration of Dulanermin
Description: The dulanermin serum concentration was measured using enzyme linked immunosorbent assay (ELISA).
Time Frame: Blood samples were taken 0.5, 1.5, 2, 3, 5, 7 and 24 hours after the start of the infusion on Day 1 of Cycle 1.
Population: Safety-evaluable population
Measure: Mean (Standard Deviation); unit: µg/ml
Groups:
- Phase Ib Dulanermin: Participants received 4.0 mg/kg/day or 8.0 mg/kg/day dose of dulanermin, administered by intravenous (IV) infusion for 5 consecutive days at the start of each 21-day treatment cycle for up to four cycles. Participants also received rituximab administered by IV infusion at 375 mg/m^2 weekly for up to eight doses.
- Phase II Dulanermin: Participants received 8.0 mg/kg/day dose of dulanermin, administered by intravenous (IV) infusion for 5 consecutive days at the start of each 21-day treatment cycle for up to four cycles. Participants may also have received rituximab administered by IV infusion at 375 mg/m^2 weekly for up to eight doses.
Arm/Group | Phase Ib Dulanermin | Phase II Dulanermin
Number analyzed (Participants) | 12 | 43
µg/ml
  30 minutes after the start of infusion | 0.109 (0.37) | 0.001 (0.00)
  1.5 hours after the start of infusion | 40.4 (19.03) | 51.5 (14.00)
  2 hours after the start of infusion | 49.9 (32.04) | 79.8 (22.54)
  3 hours after the start of infusion | 29.5 (20.75) | 28.7 (10.13)
  5 hours after the start of infusion | 2.21 (1.87) | 9.89 (21.86)
  7 hours after the start of infusion | 4.89 (15.69) | 0.445 (0.26)
  24 hours after the start of infusion | 0.324 (0.66) | 0.002 (0.00)

ADVERSE EVENTS:
Time Frame: Adverse events occurring on or after the first treatment through Study Termination (up to approximately 13 months for phase Ib and up to approximately 33 months for phase II) are summarized.
Description: Evaluation is on all Treated Patients.
Arm/Group | Phase Ib - Dulanermin 4 mg/kg | Phase Ib - Dulanermin 8 mg/kg | Phase II - Rituximab | Phase II - Combination Therapy | Phase II - Dulanermin
Serious Adverse Events (participants affected / at risk) | 1/6 | 1/6 | 1/22 | 4/26 | 0/11
Other Adverse Events (participants affected / at risk) | 6/6 | 6/6 | 16/22 | 22/26 | 8/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase Ib - Dulanermin 4 mg/kg (N=6) | Phase Ib - Dulanermin 8 mg/kg (N=6) | Phase II - Rituximab (N=22) | Phase II - Combination Therapy (N=26) | Phase II - Dulanermin (N=11)
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
CONSTIPATION (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
INFUSION RELATED REACTION (General disorders) | 0 | 0 | 0 | 1 | 0
PNEUMONIA (Infections and infestations) | 0 | 0 | 0 | 1 | 0
MYELODYSPLASTIC SYNDROME (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
ILEUS PARALYTIC (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
SEPSIS (Infections and infestations) | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phase Ib - Dulanermin 4 mg/kg (N=6) | Phase Ib - Dulanermin 8 mg/kg (N=6) | Phase II - Rituximab (N=22) | Phase II - Combination Therapy (N=26) | Phase II - Dulanermin (N=11)
DIARRHOEA (Gastrointestinal disorders) | 2 | 2 | 2 | 2 | 0
NAUSEA (Gastrointestinal disorders) | 2 | 2 | 4 | 4 | 0
VOMITING (Gastrointestinal disorders) | 2 | 1 | 3 | 3 | 0
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 2 | 0 | 0 | 1 | 0
CONSTIPATION (Gastrointestinal disorders) | 0 | 2 | 1 | 4 | 0
ABDOMINAL DISCOMFORT (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
DYSPHAGIA (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
ORAL PAIN (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
SENSITIVITY OF TEETH (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
STOMATITIS (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
TOOTHACHE (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 | 0 | 2 | 2 | 0
HAEMORRHOIDS (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
FATIGUE (General disorders) | 6 | 3 | 2 | 3 | 3
CHILLS (General disorders) | 1 | 3 | 0 | 0 | 0
PYREXIA (General disorders) | 2 | 1 | 0 | 5 | 0
CATHETER SITE PAIN (General disorders) | 2 | 0 | 0 | 0 | 0
CHEST PAIN (General disorders) | 2 | 0 | 1 | 1 | 0
CATHETER SITE ERYTHEMA (General disorders) | 1 | 0 | 0 | 0 | 0
CATHETER SITE PRURITUS (General disorders) | 1 | 0 | 0 | 0 | 0
FEELING COLD (General disorders) | 1 | 0 | 0 | 0 | 0
GAIT DISTURBANCE (General disorders) | 0 | 1 | 0 | 0 | 0
MUCOSAL INFLAMMATION (General disorders) | 1 | 0 | 0 | 0 | 0
OEDEMA PERIPHERAL (General disorders) | 1 | 0 | 0 | 1 | 0
PAIN (General disorders) | 0 | 1 | 1 | 1 | 0
SWELLING (General disorders) | 0 | 1 | 0 | 0 | 0
ASTHENIA (General disorders) | 0 | 0 | 0 | 4 | 2
HERNIA (General disorders) | 0 | 0 | 0 | 0 | 1
RASH (Skin and subcutaneous tissue disorders) | 2 | 3 | 2 | 0 | 0
NIGHT SWEATS (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0 | 0
PRURITUS (Skin and subcutaneous tissue disorders) | 1 | 1 | 2 | 0 | 0
DRY SKIN (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
EXFOLIATIVE RASH (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
HYPERHIDROSIS (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
SKIN INDURATION (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
DECREASED APPETITE (Metabolism and nutrition disorders) | 3 | 1 | 2 | 0 | 0
HYPERKALAEMIA (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
HYPOMAGNESAEMIA (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
METABOLIC ACIDOSIS (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
FLUID RETENTION (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
HEADACHE (Nervous system disorders) | 1 | 1 | 1 | 4 | 0
PARAESTHESIA (Nervous system disorders) | 0 | 2 | 0 | 0 | 0
SINUS HEADACHE (Nervous system disorders) | 0 | 2 | 0 | 0 | 0
TREMOR (Nervous system disorders) | 1 | 1 | 0 | 0 | 0
DIZZINESS (Nervous system disorders) | 0 | 1 | 1 | 0 | 1
DYSGEUSIA (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
HYPOGEUSIA (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
NEUROPATHY PERIPHERAL (Nervous system disorders) | 0 | 0 | 0 | 2 | 0
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 3 | 1 | 0
COUGH (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 3 | 2 | 0
SINUS CONGESTION (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 2 | 1
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
LUNG CONSOLIDATION (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
PRODUCTIVE COUGH (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 1 | 0
RESPIRATORY DISTRESS (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
RESPIRATORY TRACT CONGESTION (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
RHINORRHOEA (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 0
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 3 | 0 | 4 | 0 | 0
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 2 | 0
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 0
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 2 | 0 | 0 | 0 | 0
GROIN INFECTION (Infections and infestations) | 1 | 0 | 0 | 0 | 0
HERPES ZOSTER (Infections and infestations) | 1 | 0 | 1 | 0 | 0
PNEUMONIA (Infections and infestations) | 1 | 0 | 0 | 0 | 0
ORAL HERPES (Infections and infestations) | 0 | 0 | 1 | 4 | 0
VIRAL INFECTION (Infections and infestations) | 0 | 0 | 0 | 0 | 2
RHINITIS (Infections and infestations) | 0 | 0 | 0 | 0 | 1
LIPASE INCREASED (Investigations) | 1 | 1 | 0 | 0 | 0
BACTERIAL TEST POSITIVE (Investigations) | 1 | 0 | 0 | 0 | 0
BLOOD AMYLASE INCREASED (Investigations) | 0 | 1 | 0 | 0 | 0
DEEP VEIN THROMBOSIS (Vascular disorders) | 0 | 1 | 0 | 0 | 0
HYPOTENSION (Vascular disorders) | 1 | 0 | 0 | 0 | 0
PHLEBITIS SUPERFICIAL (Vascular disorders) | 1 | 0 | 0 | 0 | 0
HYPERTENSION (Vascular disorders) | 0 | 0 | 1 | 1 | 1
PHLEBITIS (Vascular disorders) | 0 | 0 | 0 | 2 | 0
ANXIETY (Psychiatric disorders) | 0 | 1 | 1 | 0 | 0
INSOMNIA (Psychiatric disorders) | 1 | 0 | 1 | 0 | 0
NERVOUSNESS (Psychiatric disorders) | 0 | 1 | 1 | 0 | 0
NOCTURIA (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
RENAL FAILURE ACUTE (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
ANAEMIA (Blood and lymphatic system disorders) | 1 | 0 | 1 | 0 | 0
COAGULOPATHY (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0
DISSEMINATED INTRAVASCULAR COAGULATION (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0
NEUTROPENIA (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 1 | 0 | 1 | 0 | 0
LEFT VENTRICULAR DYSFUNCTION (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
RIGHT VENTRICULAR DYSFUNCTION (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
DEAFNESS UNILATERAL (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0
ADRENAL INSUFFICIENCY (Endocrine disorders) | 1 | 0 | 0 | 0 | 0
DRY EYE (Eye disorders) | 0 | 1 | 0 | 0 | 0
VISION BLURRED (Eye disorders) | 0 | 0 | 0 | 1 | 1
HEPATIC FAILURE (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0
CONTUSION (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0 | 0
INCISION SITE PAIN (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
DRUG HYPERSENSITIVITY (Immune system disorders) | 0 | 0 | 0 | 2 | 0

LIMITATIONS AND CAVEATS:
The Sponsor terminated the study on 5 May 2010, prior to the completion of the 36-month follow-up (FU) period, based on the primary analysis results. All patients were off-study or in survival FU (the treatment period was completed).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.